CLINICAL TRIAL: NCT02694146
Title: Clinical Trial Randomized, Double-blind Controlled, Phase III, to Evaluate the Use of Platelet Rich Plasma in Front Hyaluronic Acid in Coxarthrosis
Brief Title: Clinical Trial to Evaluate the Use of Platelet Rich Plasma in Front Hyaluronic Acid in Coxarthrosis
Acronym: COX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COX1985; 2014-004120-21 (EudraCT Number)
Record Dates: First submitted 2016-02-09; First posted 2016-02-29 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2017-05

CONDITIONS: Coxarthrosis
Keywords: platelet-rich plasma (PRP); hyaluronic acid (Hylan G-F 20).; NSAIDs; WOMAC
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — hylan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP (platelet rich plasma) (Experimental): 37 patients with coxarthrosis are treated with 6ml of PRP (platelet rich plasma), obtained from blood extracted from patients in the 20 minutes prior to infiltration thereof.
  For PRP administration:
  * The injection should be performed at room temperature.
  * The administration should be carried out under aseptic conditions.
  * The patient will be placed in the supine position and the administration will be performed by an anterolateral approach.
  * The PRP is injected into the synovial space.
  Interventions: Drug: Platelet rich plasma
- Hylan G-F 20 (Synvisc-One ®) (Active Comparator): 37 patients with coxarthrosis are treated with a pre-filled syringe of hyaluronic acid 60mg / 6ml (Synvisc-One ®).
  It is necessary to remove synovial fluid before injecting Hylan G-F 20.
  * The injection should be performed at room temperature.
  * The administration should be carried out under aseptic conditions.
  * The patient will be placed in the supine position and the administration will be performed by an anterolateral approach.
  * The Hylan G-F 20 is injected into the synovial space.
  * After injecting Hylan G-F 20 the patient should stand 5 minutes.
  Interventions: Drug: Hylan G-F 20

INTERVENTIONS:
Drug: Platelet rich plasma — Platelet rich plasma (PRP) is a platelet concentrated obtained from autologous blood centrifugation. This concentration technique provides larger amounts of biologically active molecules, mainly growth factors that are responsible for tissue repair. PRP (platelet rich plasma) contains a higher concentration of platelets from baseline (150,000-350,000 / ul).
  Other Names: PRP
  Arms: PRP (platelet rich plasma)
Drug: Hylan G-F 20 — Hylan G-F 20 is a viscous, sterile and non-pyrogenic elasto fluid containing hylan. Hylans are byproducts from hyaluronate (hyaluronic acid sodium salt), consisting of repeating disaccharides of N-acetylglucosamine and sodium glucuronate. Hylan G-F 20 replaces and supplements the synovial fluid. It is effective at any stage of the joint pathology.
  Other Names: Synvisc-One
  Arms: Hylan G-F 20 (Synvisc-One ®)

SUMMARY:
To evaluate the efficacy and safety of platelet rich plasma (PRP) in patients with coxarthrosis who don´t respond to treatment with NSAIDs, compared to treatment with hyaluronic acid (Hylan G-F 20).

ELIGIBILITY:
Inclusion Criteria:

* Patients> 30 years.
* Patients who voluntarily express their intention to participate by informed consent.
* Diagnosis of coxarthrosis who have failed conservative treatments for 6 months
* Women of childbearing potential must have a negative pregnancy test during screening and must agree to use adequate contraception (or two contraceptive methods, of which one is barrier) while participating in the trial.

Exclusion Criteria:

* Treatment with infiltrations 3 months prior to the study
* Prior treatment with NSAIDs 24h prior to extraction
* Pre-Surgical Treatment of Hip affects
* Diabetics
* Severe liver or kidney disease at the time of extraction
* Thrombocytopenia (<100,000 platelets / ml) at baseline
* Anemia (Hb 9 <mg / dl) at baseline
* Hyaluronic acid Allergy
* History crystal arthropathy, inflammatory arthritis or neuropathic arthropathy.
* Acetabular protrusions
* History of infectious arthritis
* Excessive deformity (acetabular dysplasia, Perthes)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
EVA scale for pain measure. | Through study completion, an average of 1 year.
  The patient assesses the sensation of pain following a horizontal visual analog scale (EVA) with values between 0 ("no pain") and the value 100 ("excruciating pain"). The records taken are recorded in the medical record of the patient.
Harris Hip Score for pain, function and range of motion measure. | Through study completion, an average of 1 year.
  It is a questionnaire developed to evaluate hip surgery or replacement. It is widely used for evaluation of hip disorders and treatment methods.
WOMAC questionnaire for pain, stiffness and joint mobility measure. | Through study completion, an average of 1 year.
  It is a standardized questionnaire, widely used for assessment of both knee and hip osteoarthritis. It consists of five items for assessing pain (range 0-20), two items that assess the stiffness (range 0-8) and 17 items that evaluate the functionality of the joint (range 0-68).

OTHER OUTCOMES:
Adverse events. | Through study completion, an average of 1 year.
  All adverse events (AEs) are recorded in the case report data from the time that the patient sign the informed consent, indicating the nature of adverse events and their description in both: the experimental group and the comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Javier Roca Ruiz, Graduate, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (2):
- Spain (2):
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario Virgen Macarena, Seville